CLINICAL TRIAL: NCT07400705
Title: Short-term Outcomes of High Tibial Osteotomy Using a Plate Versus a Plate With an Interbody Fusion Cage in Adolescent Tibia Vara : a Comparative Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Atef Ahmed Hafez, resident doctor in sohag orthopedic department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-26-1-3MS
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Tibia Vara in Children
Keywords: Tibia vara is a progressive angular deformity of the lower limb centered at the proximal tibial physis, producing a characteristic bowing of the leg.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Corrective HTO with plate fixation only. (Active Comparator)
  Interventions: Procedure: high tibial osteotomy using interbody fusion cage
- Group B: Corrective HTO with plate fixation plus an interbody fusion cage. (Active Comparator)
  Interventions: Procedure: high tibial osteotomy using interbody fusion cage

INTERVENTIONS:
Procedure: high tibial osteotomy using interbody fusion cage — correction of adolescent tibia vara with high tibial osteotomy using interbody fusion cage

SUMMARY:
Tibia vara is a progressive angular deformity of the lower limb centered at the proximal tibial physis, producing a characteristic bowing of the leg. The condition is believed to result from an abnormal distribution of biomechanical stresses combined with an underlying genetic predisposition. (1) Excessive mechanical loading on the medial portion of the proximal tibial growth plate leads to asymmetric physeal activity, ultimately causing a pathologic varus deformity of the tibia.(²)

DETAILED DESCRIPTION:
The adolescent tibia vara may affect one or both limbs and is typically identified during or shortly before the pubertal growth spurt. (1) It is more frequently reported among individuals of African descent and those with a body mass index (BMI) greater than 40. (2) The increased body weight in these patients accentuates compressive forces on the posteromedial aspect of the proximal tibial physis,(3) resulting in localized inhibition of growth according to the Heuter-Volkmann principle, and leading to progressive varus deformity.(4) In many cases, associated deformities may also be observed at the distal tibia or femur, presenting as either varus or valgus alignment abnormalities.(5) Given the mechanical and structural nature of this deformity, corrective high tibial osteotomy (HTO) remains the cornerstone of surgical management in adolescent tibia vara. Modern fixation methods particularly the use of plate fixation versus plate combined with interbody fusion cage are being explored to enhance alignment correction, stability, and long-term outcomes in this challenging age group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged [10-18] years diagnosed with tibia vara.
* Symptomatic varus deformity centered at the proximal tibia requiring surgical correction.
* Both sexes included
* Open or transitional growth plates are suitable for HTO.

Exclusion Criteria:

* Prior tibial realignment surgery on the same side.
* Ages below 10 years or above 18 years
* Active infection, progressive metabolic disorder (e.g., rickets) or skeletal dysplasia, neuromuscular disorder, or systemic inflammatory arthritis.
* Complex deformities need external fixation as the first-line treatment.
* Patients with chronic comorbidities.
* Associated with fractures in the same limb

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2025-10-06 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2026-10-06 (Estimated)

PRIMARY OUTCOMES:
correction of tibia vara radiologically | 6 months
  Change in MPTA from baseline to 6 months, measured on radiographs by two blinded observers.
correction of tibia vara on radiographs | 6 months
  Change in MPTA from baseline to 6 months, measured on radiographs by two blinded observers.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Univesity Hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data and related study documents (protocol, CRF, SAP) will be made available upon reasonable request. Data will be accessible starting 6 months after the main results publication and will remain available for at least 5 years. Access will be granted to qualified researchers after approval of a research proposal and completion of a data sharing agreement. Data will be stored in a secure, publicly accessible repository
Supporting Information: SAP
Time Frame: 6 months anf for 5 years

REFERENCES:
- [Background] Jang SH, Chang CH, Jung YJ, Kwon HG. Hypersomnia due to injury of the ventral ascending reticular activating system following cerebellar herniation: A case report. Medicine (Baltimore). 2017 Jan;96(1):e5678. doi: 10.1097/MD.0000000000005678. PMID 28072702
- See also: Anteromedial incision , osteotomy cut and open using laminar spreader then insert suitable size cage and apply plate — https://www.orthobullets.com/recon/3135/high-tibial-osteotomy